CLINICAL TRIAL: NCT05622656
Title: Intraperitoneal Installation of Can Enhance Postoperative Analgesia of Caesarean Section
Brief Title: Dexmedetomidine Reduce Postoperative Pain of C-section
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First People's Hospital of Chenzhou (Other)
Responsible Party: Principal Investigator, zhiming zhang, MD, Ph.D, First People's Hospital of Chenzhou
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 202002
Record Dates: First submitted 2022-11-12; First posted 2022-11-18 (Actual); Last update posted 2022-11-18 (Actual); Status verified 2022-11

CONDITIONS: Pain, Postoperative
Keywords: Intraperitoneal spraying; Dexmedetomidine; Cesarean section; Postoperative analgesia
MeSH Terms: conditions — Pain, Postoperative | interventions — Dexmedetomidine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Intraperitoneal instillation of normal saline
  Interventions: Drug: Placebo
- Dexmedetomidines (Active Comparator): Intraperitoneal instillation Dexmedetomidine 5ug/ml (10ml,50ug)
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine 0.0005%
  Other Names: Dexmedetomidine Hydrochloride
  Arms: Dexmedetomidines
Drug: Placebo — 0.9% Sodium Chloride Solution
  Other Names: Normal saline
  Arms: Placebo

SUMMARY:
The purpose of this study was to make sure whether the infiltration of dexmedetomidine around the uterus can reduce the pain of cesarean section surgery.Studies have shown that the use of local anesthetic infiltration around the uterus can reduce pain after cesarean section surgery.In observed group, 50ug of dexmedetomidine (volume 10ml) was infiltrated around the uterus at the end of the caesarean section, while in controled group, 10ml normal saline as placebo was infiltrated around the uterus. VASs was accessed in 2h 12h,24h,48h after surgery.

DETAILED DESCRIPTION:
Cesarean section is one of the most common inpatient surgical procedures in the world, and in China, with the implementation of the comprehensive two-child policy, the number of elderly mothers and patients undergoing another cesarean section has gradually increased, and the cesarean section rate has also gradually increased; however, despite the many measures taken to control post-cesarean pain, there are still many people with inadequate pain control. Pain after cesarean delivery can have a significant negative impact on both the physical and psychological aspects of the mother and lead to complications such as thromboembolism, chronic pain and depression. Currently, a variety of methods are available to relieve post-cesarean pain, such as patient controlled intravenous analgesia (PCIA), patient controlled epidural analgesia (PCEA), transversus abdominis plane block (TAPB), etc. However, these analgesic methods are not perfect, and each has its own shortcomings. The currently prevalent ERAS concept focuses on multimodal analgesia and minimizing the use of opioids to reduce perioperative stress and reduce opioid nociceptive allergy. Compared to the technical difficulties, risks and other potential complications, abdominal medication has some advantages.

Intraperitoneal spray of local anesthetic (IPLA) has become a commonly used method of analgesia after laparotomy. Intraperitoneal administration is simple, safe, and can relieve postoperative pain, shorten the length of hospital stay, and improve comfort.

One study showed that the use of intraperitoneal infusion of lidocaine (400 mg) improved pain management in the early postoperative period after cesarean section and reduced the number of patients requiring systemic opioids in the immediate postpartum period. It has also been demonstrated that in patients undergoing bariatric surgery, intraoperative intraperitoneal spraying of ropivacaine resulted in effective postoperative pain relief, less need for morphine postoperatively, earlier activity and feeding, and shorter hospital stays, that effective pain control encouraged early bedtime, reduced the risk of thrombosis, and reduced pulmonary complications such as atelectasis or pneumonia, and that 24-hour postoperative blood counts showed significantly lower leukocyte counts were significantly lower.

Dexmedetomidine is a potent, multifunctional, highly selective α2-adrenergic agonist. It has been shown in the literature that the application of dexmedetomidine can effectively reduce the perioperative stress response, significantly reduce the dosage of opioids in the perioperative period and prevent the transformation of acute postoperative pain into chronic pain. Some animal experiments have shown that dexmedetomidine alone has obvious analgesic effect when sprayed intraperitoneally with 12.5μg/kg of dexmedetomidine, the peak time is 20-30 minutes after administration, and the duration of action is 90 minutes. There are few studies on the use of dexmedetomidine alone intraperitoneally to reduce postoperative pain in the clinical setting and there is a lack of data to support its use in post-caesarean pain.

The purpose of this study was to assess the effect of intraperitoneal dexmedetomidine 50μg at the end of cesarean delivery on maternal pain scores and satisfaction in the context of a multimodal analgesic protocol.

The investigators hypothesized that intraperitoneal dexmedetomidine would reduce VAS pain scores, reduce the number of patient-administered intravenous analgesic pump uses and opioid-related side effects, and increase maternal satisfaction after cesarean delivery.

ELIGIBILITY:
Inclusion Criteria:

* ASA Ⅰ or Ⅱ patients
* 18-50 years of age
* BMI<40
* Term pregnancy
* Singleton pregnancy
* Spinal anesthetic
* Patients who have given pre-operative informed written consent

Exclusion Criteria:

* Patients who refuse or are unable to give consent
* ASA>Ⅱ
* Multiple gestation
* Chronic pain
* allergic to any medication in the study protocol

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Pain Score (VAS) 48hr rest | 48 hours
  VAS score (VAS 0-10 cm) for maternal pain on rest at 48 hours postcesarean delivery
Pain Score (VAS) 48hr movement | 48 hours
  VAS score (VAS 0-10 cm) for maternal pain on movement at 48 hours postcesarean delivery

SECONDARY OUTCOMES:
Pain Score (VAS) 2hr rest | 2 hours
  VAS score (VAS 0-10 cm) for maternal pain on rest at 2 hours postcesarean delivery
Pain Score (VAS) 2hr movement | 2 hours
  VAS score (VAS 0-10 cm) for maternal pain on movement at 2 hours postcesarean delivery
Pain Score (VAS) 24hr rest | 24 hours
  VAS score (VAS 0-10 cm) for maternal pain on rest at 24 hours postcesarean delivery
Pain Score (VAS) 24hr movement | 24 hours
  VAS score (VAS 0-10 cm) for maternal pain on movement at 24 hours postcesarean delivery
Effective presses of PCIA pump 48hrs | 48 hours
  Number of effective presses of PCIA pump at 48 hours postcesarean delivery
Patient satisfaction 48hrs | 48 hours
  Patient satisfaction at 48 hours postcesarean
Bowel function | 48 hours
  Return of bowel function as assessed by passing flatus
Side Effect scores | 48 hours
  Nausea, vomiting and pruritis score at 24 hours and 48 hours postcesarean delivery
Flurbiprofen Axetil consumption 48hrs | 48 hours
  Flurbiprofen Axetil consumption within 48 hours postcesarean delivery

CONTACTS AND LOCATIONS:
Locations (1):
- Zhiming Zhang, Chenzhou, Hunan, China